CLINICAL TRIAL: NCT02071888
Title: A Phase 1 Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Escalating Oral Doses of the Glutaminase Inhibitor CB-839 in Patients With Advanced and/or Treatment-Refractory Hematological Malignancies
Brief Title: Study of the Glutaminase Inhibitor CB-839 in Hematological Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-002
Record Dates: First submitted 2014-02-14; First posted 2014-02-26 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Non-Hodgkin's Lymphoma (NHL); Multiple Myeloma; Waldenstrom's Macroglobulinemia (WM); Other B-cell NHL Subtypes, Including WM; T-cell NHL
Keywords: Non-Hodgkin's lymphoma; Waldenstrom's macroglobulinemia; Multiple myeloma; glutaminase; glutamine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — CB-839; Dexamethasone; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CB-839 (Experimental): CB-839 is administered as oral capsules three times daily (TID) or twice daily with food (BIDf) in 21-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839
- CB-839 and low dose dexamethasone (Experimental): CB-839 is administered as oral capsules twice daily with food (BIDf) in 28 day cycles in combination with dexamethasone until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: CB-839 and low dose dexamethasone
- CB-839, pomalidomide, and low dose dexamethasone (Experimental): CB-839 is administered as oral capsules twice daily with food (BIDf) in 28 day cycles in combination with pomalidomide and dexamethasone until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: CB-839 and low dose dexamethasone; Drug: CB-839, pomalidomide, and low dose dexamethasone

INTERVENTIONS:
Drug: CB-839 — Glutaminase inhibitor
Drug: CB-839 and low dose dexamethasone — CB-839 and low dose dexamethasone
  Other Names: CBd
  Arms: CB-839 and low dose dexamethasone; CB-839, pomalidomide, and low dose dexamethasone
Drug: CB-839, pomalidomide, and low dose dexamethasone — CB-839, pomalidomide, and low dose dexamethasone
  Other Names: CBPd
  Arms: CB-839, pomalidomide, and low dose dexamethasone

SUMMARY:
Many tumor cells, in contrast to normal cells, have been shown to require the amino acid glutamine to produce energy for growth and survival. To exploit the dependence of tumors on glutamine, CB-839, a potent and selective inhibitor of the first enzyme in glutamine utilization, glutaminase, will be tested in this Phase 1 study in patients with advanced hematologic malignancies.

This study is an open-label Phase 1 evaluation of CB-839 in subjects with hematological tumors. Patients will receive CB-839 capsules orally two or three times daily. The study will be conducted in 2 parts. Part 1 is a dose escalation study to identify the recommended Phase 2 dose and will enroll patients with advanced and/or treatment-refractory Non-Hodgkin's Lymphoma (NHL), Multiple Myeloma (MM), or Waldenström's macroglobulinemia (WM)

In Part 2, all patients will receive the recommended Phase 2 dose. This part will enroll patients with advanced and/or treatment-refractory Non-Hodgkin's Lymphoma (NHL), Multiple Myeloma (MM), or Waldenström's macroglobulinemia (WM). All patients will be assessed for safety, pharmacokinetics (plasma concentration of drug), pharmacodynamics (inhibition of glutaminase), biomarkers (biochemical markers that may predict responsiveness in later studies), and tumor response.

As an extension of Part 2, a cohort of patients with relapsed and refractory MM will be enrolled to receive low dose dexamethasone and CB-839. A second cohort of patients with relapsed or refractory disease following at least 2 prior treatment regimens will be enrolled to receive CB-839 in combination with standard-dose pomalidomide and low-dose dexamethasone to further evaluate this triple combination.

ELIGIBILITY:
Disease-Specific Inclusion Criteria

Patients must have one of the following diseases that is either relapsed or refractory to 2 or more prior treatments:

* NHL: At least one measurable lesion
* WM: Measurable IgM, with a minimum level of ≥ 2x ULN
* MM: Serum M-protein ≥ 0.5 g/dL and/or urine M-protein ≥ 200 mg/24 hr. In Part 2, disease that is considered measurable per the IMWG criteria

Other Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life Expectancy of at least 3 months
* Adequate hepatic, renal, cardiac and hematological function

Exclusion Criteria

* Any other current malignancy
* Treatment with an unapproved, investigational therapeutic agent, immunotherapy or biological therapy within 21 days prior to the first dose of study drug
* Recent bone marrow transplant
* Unable to receive medications by mouth
* Major surgery within 28 days before the first dose of study drug
* Uncontrolled, active infection; patients who are known to have HIV infection/ seropositivity, Hepatitis A, B, or C, or CMV reactivation
* Significant neurotoxicity/neuropathy (Grade 3 or higher) within 14 days prior to the first dose of study drug
* Refractory nausea and vomiting or other situation that may preclude adequate absorption
* Other conditions that could interfere with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CB-839: Incidence of adverse events | Every 21 days from study start until disease progression or unacceptable toxicity, assessed for an expected average of 6 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the Curve (AUC) of CB-839 concentration in blood | Study Days 1, 15, and 22
Pharmacodynamics: % inhibition of glutaminase in blood | Study Days 1 and 15
Clinical activity: Change in tumor size from baseline | Every 9 weeks (NHL) or 3 weeks (MM and WM), assessed for an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Orford, MD, PhD, Study Director — Calithera Biosciences
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Winship Cancer Institute of Emory School of Medicine, Atlanta, Georgia
  - John Theruer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee